CLINICAL TRIAL: NCT01313975
Title: Disturbances of the Sodium and Fluid Balance in Patients With Severe Traumatic Brain Injury and Non-traumatic Subarachnoid Hemorrhage. A Systematic Observational Study
Brief Title: Electrolyte and Fluid Disturbances in Subarachnoid Hemorrhage and Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Foundation for research in Anaesthesie and Intensive Care Medicine (Unknown); Brahms AG (Industry)
Responsible Party: Jan Wiegand, MD, Department of Intensive Care Medicine University Hospital Bern, Switzerland
Other Study IDs: 203/10
Record Dates: First submitted 2011-02-21; First posted 2011-03-14 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Electrolyte Disturbances; Subarachnoid Hemorrhage; Traumatic Brain Injury; Natriuretic Peptides
Keywords: Electrolyte disturbances; Fluid balance; subarachnoid hemorrhage; traumatic brain injury; Cerebral salt wasting; SIADH; Diabetes insipidus
MeSH Terms: conditions — Subarachnoid Hemorrhage; Brain Injuries, Traumatic; Inappropriate ADH Syndrome; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with non-traumatic subarachnoid hemorrhage
- 2: Patients with severe traumatic brain injury

SUMMARY:
During the course of their acute illness patients with subarachnoid hemorrhage and severe traumatic brain injury often develop disturbances in their fluid balance and electrolyte homeostasis. These shifts are associated with worse outcome and increased morbidity.

The aim of this observational study is to systematically analyze the incidence, characteristics, potential diagnostic markers and predisposing factors of such disturbances. The investigators hypothesize that many disturbances cannot be classified with a standard diagnostic approach and that variable fluid management contributes to their pathophysiology.

Patients will be closely monitored clinically and the exact fluid and electrolyte balances will be recorded. Treatment decisions are within the bedside physicians responsibility. Baseline fluid management is standardised. No interventions are planned. The observation period equal the duration of ICU stay.

DETAILED DESCRIPTION:
Background

Electrolyte disturbances and fluid shifts are common in patients with subarachnoid hemorrhage (SAH) or traumatic brain injury (TBI). They usually have a rapid onset with impact on morbidity (possibly mortality) and length of stay. So far the understanding of underlying pathophysiologies and the contribution of iatrogenic influences is not fully understood.

Only limited evidence and data on classification, management and outcome of patients exists.

Objective

To describe the incidence, characteristics and duration of sodium and fluid disturbances in patients with SAH or TBI.

To document exact fluid and electrolyte management To evaluate predisposing factors and potential predicting biomarkers such as natriuretic peptides, renin-aldosterone system.

Methods

Prospective systematic observational study with 50 patients in the SAH group and 50 patients in the TBI group.

8hourly clinical assessment, blood and urin samples. Defined trigger points for additional measurements.

Continuous fluid balance documentation Daily measurement of natriuretic peptides, aldosterone and renin

ELIGIBILITY:
Inclusion Criteria:

* non-traumatic subarachnoid hemorrhage
* severe traumatic brain injury (GCS<9)

Exclusion Criteria

* younger than 18 years
* time to admission after injury or bleed more than 7days
* death expected in less than 12hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intenisve Care Medicine patients with non-traumatic subarachnoid hemorrhage or severe traumatic brain injury
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Incidence of sodium-fluid disturbances | 14 days

SECONDARY OUTCOMES:
Type of sodium abnormality | 14 days
Haemodynamic changes, 8hourly urine output, 8hourly fluid and sodium balance, changes in fluid management by treating doctors associated with sodium disturbances | 14 days
  We measure all parameters for multivariate analysis to find common predictors for sodium and fluid balance disturbances in these patients
Associated changes in natriuretic peptide levels | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Jan Wiegand, MD, Principal Investigator — Dep. Intensive Care Medicine, University Hospitals Bern; Stephan Jakob, MD, PhD, Study Director — Dep. Intensive Care Medicine, University Hospitals Bern; Jukka Takala, MD PhD, Study Chair — Dep. Intensive Care Medicine, University Hospitals Bern
Locations (1):
- Dep. of Intensive Care Medicine Bern University Hospital, Bern, Switzerland